CLINICAL TRIAL: NCT05284071
Title: Actiste® Diabetes Management as a Service (ADMS) - A Clinial Investigation With Insulin Treated Diabetes Patients in the UK
Brief Title: Actiste® Diabetes Management as a Service (ADMS) Clinical Investigation
Acronym: ADMSUK01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Care Alliance NHS Foundation Trust (Other)
Collaborators: Brighter AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S21DIAB02-S
Record Dates: First submitted 2022-02-22; First posted 2022-03-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Diabetes type1; Diabetes type2
Keywords: Diabetes Management; HbA1c; Patient; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Single-Arm (Experimental): This is a prospective, single-arm, post-market study to verify clinical performance, treatment satisfaction and adherence, and safety of Actiste 1.0 (Actiste) and the Companion app with TBL Backend when used as intended by subjects diagnosed with T1DM or T2DM.
  Interventions: Device: Device: Actiste 1.0 and the Companion app with TBL Backend

INTERVENTIONS:
Device: Device: Actiste 1.0 and the Companion app with TBL Backend — Actiste automatically logs and shares real-life data on blood glucose values and actual injected insulin doses. With Actiste's built-in sensor, the exact injected dose is displayed and saved in the device memory together with a time stamp, which makes it easy for the user to know how much and when the insulin was injected, and spot missed doses. This simplifies the daily diabetes care for the user and thus may improve the quality of life for people with diabetes and may improve the patients' adherence to treatment plans. Actiste automatically logs and shares real-life data on blood glucose values and actual injected insulin doses. With Actiste's built-in sensor, the exact injected dose is displayed and saved in the device memory together with a time stamp, which makes it easy for the user to know how much and when the insulin was injected, and spot missed doses. This simplifies the daily diabetes care for the user and thus may improve the quality of life for people with diabetes.

SUMMARY:
The overall aim of the clinical investigation is to confirm clinical performance, treatment satisfaction, adherence and safety of Actiste 1.0 and the Companion

- Page 1 of 5 - app with TBL Backend when used by subjects with diabetes in need of insulin treatment.

Primary objective:

To assess diabetes treatment satisfaction in subjects with diabetes type 1 or type 2 in need of insulin treatment when using Actiste 1.0 and the Companion app with TBL Backend

Secondary objective:

To assess clinical performance and treatment adherence in subjects with diabetes type 1 or type 2 in need of insulin treatment when using Actiste 1.0 and the Companion app with TBL Backend

DETAILED DESCRIPTION:
This is a prospective, single-arm, post-market clinical investigation to verify clinical performance, treatment satisfaction, adherence and safety of Actiste 1.0 and the Companion app with TBL Backend, referred to as Actiste diabetes management system (ADMS) when used as intended by subjects diagnosed with Diabetes Mellitus Type 1 or Type 2 (T1DM or T2DM). In total, 70 subjects diagnosed with T1DM or T2DM (35 subjects per type) using Glargine U100 basal insulin with or without oral antidiabetic drugs/bolus insulin regimen will be enrolled at 1 site in the UK. Each subject will be evaluated during a period of 6 months. Eight (8) visits are planned for each subject during the clinical investigation, including 3 visits to the study clinic and 5 visits conducted as telephone calls. During the visits, evaluations will be performed to assess blood glucose levels, adherence to the treatment plan, quality of life and treatment satisfaction. Data on blood glucose values, insulin injections and diabetesrelated data from the Companion app and TBL Backend will be shared by the subject.Each participant will be provided with the ADMS, including Actiste 1.0, and the Companion app for their smartphone with the TBL Backend. No comparator will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Adult males and females =18 years old
3. Diagnosed with diabetes I or II, since = 6 months prior to entering the investigation, according to investigator judgement
4. Currently using insulin as a component of the diabetes therapy, Sanofi Lantus insulin (glargine U100 insulin incartridge or disposable pen)± any form or manufacturer of oral antidiabetic drugs (OADs)/bolus insulin regimen/GLP-1RA
5. HbA1c 64-86mmol/mol in the last 30 days
6. Patients using Self-Monitoring of Blood Glucose (SMBG) = 1 month prior to entering the investigation
7. Able to use smartphone (iOS or Android)independently, according to investigator judgement
8. Currently using a system compatible smartphone (Android and iOS smartphones: iOS platform versions from 12.0 to 14.x and Android platform versions from 5.1 to 11.x
9. Able to use the device independently, according to investigator judgement

Exclusion Criteria:

1. Impaired vision affecting ability to use investigation device or smartphone, according to investigator judgement
2. Patients using a flash glucose monitor, continuous glucose monitor and/ or insulin pump
3. Pregnancy or lactation at time of study participation.
4. Physical or mental impairment affecting subjects' ability to use the device, per investigator judgement
5. Person not suitable for the investigation according to the investigator judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Diabetes Treatment Satisfaction Questionnaire (change, DTSQc), at 3 months | 3 months
  The Diabetes Treatment Satisfaction Questionnaire (Change, DTSQc) will be completed during the on-site visit at 3 months. The DTSQc is a modified version of the DTSQs designed to overcome ceiling effects and to detect changes in treatment satisfaction. Answers on a 7 graded scale from -3 to 3. In majority, higher score means better outcome.

SECONDARY OUTCOMES:
Percentage and absolute change in HbA1cat 3 and 6 months, compared to baseline | 6 months
  During each on site visit, glycosylated haemoglobin(HbA1c) will be assessed. A blood sample will be taken by the site staff and HbA1c will be assessed per clinical routine at the site.
Percentage and absolute change in fasting blood glucose at 3 and 6 months, compared to baseline | 6 months
  Fasting glucose will be assessed per standard of care at the investigation site. Fasting glucose will be assessed using the Actiste device at least 4 times in the last 10 days (assessment period) before the investigation visit. The final data will be a mean of the measurements during the assessment period. The data will be extracted by the patient to a PDF file and provided to site 2 days before the visit. Site will ask what day and time the fasting blood glucose data was assessed. The data will also be summarised at the end of the investigation and the interim analysis with data from the Companion app and TBL Backend.
Absolute and percentage change in DTSQ (Status) at 6 months, compared to baseline | 6 months
  The Diabetes Treatment Satisfaction Questionnaire (Status, DTSQs) will be completed during the on-sitevisits at baseline and at 6 months.The DTSQs is recommended for measuring patient satisfaction with diabetes treatment. Answers on a 7 graded scale from 0 to 6. In majority, higher score means better outcome.
Absolute and percentage change in EQ-5D-5L (each separate question and VAS) at 3 and 6 months, compared to baseline. | 6 months
  The EQ5D5L questionnaire will be completed during the on-site visits at baseline and at 3 and 6 months. The EQ-5D-5L contains 5 questions, each with a 5 graded answer scale from "I am unable to..." to "I have no problems ...". The VAS scale is a scale from 0-100, where 100 means the best health you can imagine and 0 the worst health you can imagine
Summary of adherence in the population, from baseline to 3 months, from 3 months to end of investigation and from baseline to end of investigation. | 6 months
  Adherence will be summarised at 3 and 6 months by assessing number and percentage of missed basal insulin injections per subject during the period between the visits, compared to the subject's treatment plan. For most subjects, a basal insulin injection is performed at 22.00 in the evening, per standard clinical routine.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Heald, Dr, Principal Investigator — Northern Care Alliance NHS Foundation Trust, Stott Lane, Salford, M6 8HD
Locations (1):
- Salford Royal Hospital Northern Care Alliance NHS Foundation Trust, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No